CLINICAL TRIAL: NCT05345288
Title: Effect of Computerized Cognitive Training in Persons With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0112-22-EP
Record Dates: First submitted 2022-03-20; First posted 2022-04-25 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: The intervention group will complete the prescribed computerized cognitive training while the control group will complete the control games that are not cognitive training and offered through the BrainHQ website as well.
Who Masked: Participant
Masking Description: Participants will not know if there are in the intervention or control group until the completion of the study. The PI will know since she will have to assign the online activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Subjects randomized to the intervention group will complete prescribed cognitive training activities 3 times a week for 20-30 minutes each time for 6 weeks. Subjects randomized to the control group will complete computerized control activities that are not cognitive training on BrainHQ 3 times a week for 20-30 minutes each time for 6 weeks.
  Interventions: Device: BrainHQ cognitive training
- Control (Active Comparator): Subjects randomized to the control group will complete computerized control activities that are not cognitive training on BrainHQ 3 times a week for 20-30 minutes each time for 6 weeks.
  Interventions: Device: BrainHQ control games

INTERVENTIONS:
Device: BrainHQ cognitive training — Posit Science's BrainHQ exercises are based on the science of "neuroplasticity," also called "brain plasticity." Brain plasticity is your brain's natural ability to remodel itself throughout life. The brain is always changing, sometimes for better, and sometimes for worse. What BrainHQ's exercises do is harness that change and direct it in ways that can enhance your overall performance and improve the quality of your life. BrainHQ exercises are grouped into six categories: Attention, Memory, Brain Speed, Intelligence, People Skills, and Navigation.
  Other Names: www.brainhq.com
  Arms: Intervention
Device: BrainHQ control games — BrainHQ also offers control games for research studies. The control activities will be games similar to candy crush, connect four, gem swap and battleship.
  Other Names: www.brainhq.com
  Arms: Control

SUMMARY:
Multiple sclerosis (MS) affects approximately one million people in the United States and 2.5 million worldwide. Between one million and 1.75 million persons with MS (PwMS) worldwide are estimated to suffer from cognitive impairment. Unfortunately, there is currently no consensus on the best treatment for cognitive impairment in PwMS. The objective for this study is to determine if a computerized cognitive training using the BrainHQ platform can improve cognitive impairment in PwMS. The central hypothesis is that computerized cognitive training will show some improvement in cognitive impairment. The rationale for this study is to treat all aspects of MS, not just the physical symptoms and to help PwMS live their best life. Cognitive impairment is associated with higher rates of depression in PwMS and depression leads to medication non-adherence. This means the cognitive impairment so many PwMS are dealing with must be treated. Finding non-pharmacological interventions to mitigate cognitive declines are essential to ensure that quality of life for PwMS patients matches our ability to treat and mitigate their physical symptoms of MS. To obtain the overall objectives for this study the following specific aim will be pursued: Determine the effectiveness of computerized cognitive training on changes in cognitive impairment for PwMS. This will be accomplished by completing a randomized clinical trial with two groups: computerized cognitive training using BrainHQ and an active control group that will complete non-cognitive training programs on BrainHQ. Subjects will complete the BICAMS battery at baseline and at the end of their six week intervention. Subjects will be prescribed online activities through BrainHQ to complete 2-3 times a week for approximately 20-30 minutes each. Subjects will also be asked to wear an accelerometer for a week to determine if physical activity affects cognition. The proposed research is significant because MS is diagnosed on average at age 30, meaning a high percentage of the PwMS that are suffering with cognitive impairment are in their second, third and fourth decade when they are trying to raise a family, finish college, further their career and have active social lives.

DETAILED DESCRIPTION:
Kathy Healey, MS Specialist and participating personnel on this study, is one of the MS providers at the Nebraska Medicine MS Clinic. She helped determine the following inclusion/exclusion criteria as well as the protocol. She has enlisted the help of her colleagues to help identify eligible subjects. Patients will be identified by their MS provider as having cognitive impairment, having relapsing remitting MS, being between the ages of 19-60, not having a relapse or DMT change in the last 6 months, an EDSS of 2-5.5 and not undergoing cognitive therapy. The provider will then ask the patient if they are interested in participating in a research study and if so pass on their contact information to the PI. If patients meet the inclusion/exclusion criteria they will be asked to sign the consent form and then undergo screening to include Montreal Cognitive Assessment (MoCA), Test of Premorbid Functioning (ToPF), Generalized Anxiety Disorder (GAD-7), Beck Depression Inventory (BDI-2) and Modified Fatigue Impact Score (MFIS). While these tests are being used for screening purposed only and will not be administered by a certified neuropsychologist, if a subject answered a 2 (I would like to kill myself) or a 3 (I would kill myself if I had the chance) on the suicidal thoughts question of the BDI-II then Dr. Erica Schmidt would be contacted and the patient would be notified that the research team has to break confidentiality to help them with a safety plan that could include contacting their medical provider or sending them to the ER. Dr. Schmidt is a certified neuropsychologist and is very capable of making the proper decisions if a subject discloses moderate to high risk of suicide to ensure the safety of all subjects. If a subject answered a 1 (I have thoughts of killing myself but would not carry them out) then the subject would be asked to complete the Columbia Suicide Severity Rating Scale (C-SSRS). If the subject has more than low risk based on the C-SSRS then they would be excluded from the study and Dr. Schmidt would be contacted. All subjects that answer a one, two or three on the BDI-II will also be given a pamphlet that has information regarding how to make an appointment with a neuropsychologist as well as suicide hotline numbers.

Once screened, those who meet the inclusion criteria based on their scores will be invited to continue on in the study. Eligible participants will be randomized using a block randomization table with group assignment: computerized cognitive training or control. Dr. Wichman, a biostatistician, has created a randomization chart to use to randomly assign the subjects. Since the PI is assigning BrainHQ programs to the participants she is unblinded and can use the randomization chart.

All randomized subjects will be asked to complete the Human Activity Profile29, a physical activity questionnaire, and the Perceived Deficits Questionnaire32. They will also be asked to do a baseline Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery. The BICAMS battery consists of the Symbol Digit Modalities Test (SDMT)33, the Brief Visuospatial Memory Test Revised (BVMT-R)34 and the California Verbal Learning Test 2nd edition (CVLT-II)35. The accelerometer will be given at the enrollment visit and participants asked to wear an accelerometer during waking hours over a 7 day period. Participants will return the device to researchers by mail. This visit will take approximately two hours.

All subjects will be asked to complete the prescribed activities through BrainHQ, whether it is the control activities or the cognitive activities. Subjects randomized to the intervention group will complete prescribed cognitive training activities 3 times a week for 20-30 minutes each time for 6 weeks. Subjects randomized to the control group will complete computerized control activities that are not cognitive training on BrainHQ 3 times a week for 20-30 minutes each time for 6 weeks. The BrainHQ activities will be done on a personal computer or tablet. Subjects will not be provided devices as one of the inclusion criteria is that the patient have access to a computer and the internet. The cognitive training will consist of different exercises that are meant to improve processing speed, verbal memory and visual memory which are the domains that BICAMS tests. The control activities will be games similar to candy crush, connect four, gem swap and battleship. The subjects will be provided log in information and will not be entering any personal information on the BrainHQ application.

After 6 weeks of BrainHQ programs, subjects will return for end-of-study testing that will take approximately one hour. They will complete the BICAMS battery again as well as fill out the Perceived Deficits Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19-60 inclusive
* Expanded Disability Status Scale (EDSS) score of 2-5.5 inclusive
* Relapsing-Remitting MS according to McDonald Criteria
* 17 or above on the Montreal Cognitive Assessment (MoCA)
* 70 or above on the Test of Premorbid Functioning (TOPF)
* 29 or less on the Beck Depression Inventory (BDI-II)
* Less than 15 on the Generalized Anxiety Disorder (GAD-7)

Exclusion Criteria:

* Relapse within the last 6 months
* Disease modifying treatment (DMT) change within the last 6 months
* Primary Progressive MS or Secondary Progressive MS according to McDonald Criteria
* No access to computer/internet
* Currently undergoing treatment for cognitive impairment
* Answers a 2 or 3 on the suicidal thoughts question of the BDI-II
* Answers a 1 on the suicidal thoughts question of the BDI-II and then a Columbia Suicide Severity Rating Scale indicates more than low risk

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery | at study completion, approximately 3 months
  score change in the 3 tests that make up the BICAMS battery - Symbol Digits Modalities Test (SDMT), California Verbal Learning Test 2nd Edition (CVLT-II), Brief Visuospatial Memory Test-Revised (BVMT-R). On all 3 tests a higher score is better. The tests all have normative values and t- or z-scores to compare. Baseline and post-intervention scores will be compared to see if subjects significantly improved post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Jack, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BrainHQ website which is what the subjects will be using for the intervention and control activities. — http://www.brainhq.com